CLINICAL TRIAL: NCT05739604
Title: Serum Free Amino Acid Concentrations in Critically Ill Patients Undergoing Continuous Renal Replacement Therapy (CRRT)
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radosław Owczuk, Clinical Professor, Head of Department of Anaesthesiology and Intensive Care, Medical University of Gdansk
Other Study IDs: NKBBN/575/2019
Record Dates: First submitted 2023-02-09; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Sepsis; Amino Acid Catabolism Disorder
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Patients hospitalized in the Department of Anaesthesiology and Intensive Care with sepsis or septic shock, undergoing continuous renal replacement therapy due to acute kidney injury, in whom the outcome of treatment was survival.
  Interventions: Diagnostic Test: Blood sample analysis
- Nonsurvivors: Patients hospitalized in the Department of Anaesthesiology and Intensive Care with sepsis or septic shock, undergoing continuous renal replacement therapy due to acute kidney injury, in whom the outcome of treatment was fatal.
  Interventions: Diagnostic Test: Blood sample analysis

INTERVENTIONS:
Diagnostic Test: Blood sample analysis — The concentrations of AAs and related compounds were determined by liquid chromatography/mass spectrometry (LC/MS)

SUMMARY:
Sepsis is a life-threatening condition associated with high morbidity and mortality. The breakdown of proteins mainly from skeletal muscles leads to the release of free amino acids (FAAs). The serum FAA pool has been repeatedly assessed and found to be significantly altered in patients with sepsis/septic shock. Sepsis is well known to be the most common factor contributing to the development of acute kidney injury in critically ill patients.

The investigators want to establish the baseline profile of FAAs and their derivatives in patients with sepsis/septic shock undergoing continuous renal replacement therapy due to sepsis-associated acute kidney injury. Secondly, the investigators want to compare the FAA profiles of the survivors and nonsurvivors.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* present AKI
* requiring renal replacement therapy
* hospitalized at the ICU.

Exclusion Criteria:

* acute kidney disease requiring renal replacement therapy prior to admission to the ICU
* chronic kidney disease requiring renal replacement therapy prior to admission to the ICU
* history of past CRRT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized in ICU who met inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Evaluation the baseline profile of FAAs and their derivatives in serum in a group of patients undergoing continuous renal replacement therapy (CRRT) due to sepsis associated acute kidney injury (SA-AKI) in the Intensive care unit (ICU) | Through study completion, an average of 1 year
  Daily analysis of concentrations of amino acids (AA) and related compounds with usage of liquid chromatography/mass spectrometry (LC/MS).

SECONDARY OUTCOMES:
Comparison the free amino acids (FAA) profile of survivors and nonsurvivors | Through study completion, an average of 1 year
  Daily analysis of concentrations of amino acids (AA) and related compounds with usage of liquid chromatography/mass spectrometry (LC/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Radosław Owczuk, Prof., Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdansk - Departament of Anesthesiology and Intensive Care, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No